CLINICAL TRIAL: NCT01796990
Title: Developing a Physically More Active Lifestyle Based on One's Own Values - Randomized Controlled Trial Among Sedentary Adults
Brief Title: Developing a Physically More Active Lifestyle Based on One's Own Values - RCT Among Sedentary Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Likes - Foundation for Sport and Health Sciences (Other)
Collaborators: University of Jyvaskyla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Likes-01; LIKES-01 (Other: LIKES-01)
Record Dates: First submitted 2013-02-13; First posted 2013-02-22 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Behavior
Keywords: physical activity; psychological well-being; acceptance and commitment therapy; adults
MeSH Terms: conditions — Behavior; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- REF group (Active Comparator): The participants will get written feedback about their physical activity level after the baseline, and after 3, 6, 9 and 15 months of baseline compared to the current physical activity recommendations. Feedback will be created to illustrate participants´ activity level during the measurement week combining also the information from the diary. Feedback will be posted home and don´t include face to face interaction. As an incentive for participation, participants will also have opportunity to attend a body composition analyze and get short interpretation (15 min) of their own results in the research center.
  Interventions: Behavioral: REF
- ACT group (Other): The ACT group gets the same procedure as the REF group. In addition, they will participate the ACT based program. The intervention program consists of six group sessions, about 90 minutes per session during the 9 weeks period of time. All the participants get also pedometers for monitoring their physical activity during the intervention.
  The program aims to enhance physically active lifestyle and well-being through important life values and build committed action based on the chosen important things. The importance is also placed to a mindful awareness and flexibility to everyday actions related to physical activity. The program don´t include psycho-educational elements or counseling of the health or the health benefits of physical activity.
  Interventions: Behavioral: ACT; Behavioral: REF

INTERVENTIONS:
Behavioral: ACT — The intervention program consists of six group sessions, about 90 minutes per session during the 9 weeks period of time. The group size is about 8-10 members per one group. All the participants get also pedometers for monitoring their physical activity during the intervention.
  The program aims to enhance physically active lifestyle and well-being through important life values and build committed action based on the chosen important things. The importance is also placed to a mindful awareness and flexibility to everyday actions related to physical activity. The program don´t include psycho-educational elements or counseling of the health or the health benefits of physical activity.
  Arms: ACT group
Behavioral: REF — The participants will get written feedback about their physical activity level after the baseline, and after 3, 6, 9 and 15 months of baseline compared to the current physical activity recommendations. Feedback will be created to illustrate participants´ activity level during the measurement week combining also the information from the diary. Feedback will be posted home and don´t include face to face interaction. As an incentive for participation, participants will also have opportunity to attend a body composition analyze and get short interpretation (15 min) of their own results in the research center.

SUMMARY:
The main objective of the study is to provide data of the effectiveness and feasibility of the Acceptance and Commitment Therapy in enhancing the physically active lifestyle among sedentary adults. The psychological and motivational factors related to physical activity and behavior change will also be evaluated.

DETAILED DESCRIPTION:
In more detailed the study aimed to investigate the effectiveness of the acceptance- and commitment-based behavioural intervention concerning physical activity level and self-efficacy, as well as regarding planning and the acceptance of psychological and physical discomfort related to physical activity after 3 and 6 months compared to providing only individual written feedback on their physical activity. A further aim was to explore stability and maintenance of changes in physical activity at the 6 months follow-up. It was hypothesised that acceptance- and commitment-based behavioural intervention is more effective than feedback only in improving physical activity and related beliefs and cognitions.

ELIGIBILITY:
Inclusion Criteria:

* age 30-50 years, working status, and don´t meet the current physical activity recommendations.

Exclusion Criteria:

-

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Physical activity | baseline and change after 3, 6, 9 and 15 months
  Physical activity is measured objectively by accelerometer (Actigraph GT1M, GT3X, Actigraph, Pensacola, Florida) the last seven days.

SECONDARY OUTCOMES:
The Acceptance and Action Questionnaire, AAQ-2 | baseline and change after 3, 6, 9 and 15 months
  Psychological wellbeing is measured using the Acceptance and Action Questionnaire (AAQ-2), which is a 10-item Likert-type questionnaire that assesses people's ability to take a non-elaborative, non-judgmental approach to their internal events, so that they can focus on the present moment and act in a way that is congruent with their values and goals, rather than with their internal events (e.g., fears, urges, prejudices).
the Kentucky Inventory of Mindfulness Skills (KIMS) | baseline and change after 3, 6, 9 and 15 months
  The KIMS is a 39-item self-report inventory used to assess mindfulness skills. The questionnaire contains four different specific subscales or skills: 1) observing, 2) describing, 3) acting with awareness, and 4) accepting without judgment. Participants rated each item on a 5-point Likert type scale ranging from 1 (never or very rarely true) to 5 (almost always or always true). Items reflects either direct descriptions of the mindfulness skills or the absence of that skill, and are reverse scored.
the Beck Depression Inventory, BDI-II | baseline and change after 3, 6, 9 and 15 months
  Depressive symptoms are measured with the Beck Depression Inventory, BDI-II.
Physical activity | baseline and change after 3, 6, 9 and 15 months
  Physical activity is assessed with a questionnaire (self-reported) during the last seven days.

CONTACTS AND LOCATIONS:
Overall Officials: Anu Kangasniemi, M.Sc., Principal Investigator — Likes - Foundation for Sport and Health Sciences; Tuija Tammelin, PhD, Study Director — Likes - Foundation for Sport and Health Sciences
Locations (1):
- LIKES Foundation for Sport and Health Sciences, Jyväskylä, Finland

REFERENCES:
- [Derived] Kangasniemi AM, Lappalainen R, Kankaanpaa A, Tolvanen A, Tammelin T. Towards a physically more active lifestyle based on one's own values: the results of a randomized controlled trial among physically inactive adults. BMC Public Health. 2015 Mar 18;15:260. doi: 10.1186/s12889-015-1604-x. PMID 25848812
- [Derived] Kangasniemi AM, Lappalainen R, Kankaanpaa A, Kulmala J, Hakonen H, Tammelin T. Towards a physically more active lifestyle based on one's own values: study design of a randomized controlled trial for physically inactive adults. BMC Public Health. 2013 Jul 19;13:671. doi: 10.1186/1471-2458-13-671. PMID 23866812